CLINICAL TRIAL: NCT01632657
Title: Effect of Sumatriptan on the Postoperative Quality of Recovery After Elective Minimally Invasive Craniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Lashmi Venkatraghavan, Dr., University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-0139
Record Dates: First submitted 2012-06-28; First posted 2012-07-03 (Estimated); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Quality of Recovery; Postoperative Migrainous Headache
MeSH Terms: interventions — Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sumatriptan (Experimental): Subcutaneous injection of sumatriptan (6 mg)
  Interventions: Drug: Sumatriptan; Other: Placebo
- Placebo (Placebo Comparator): Matching placebo (0.9% saline)
  Interventions: Drug: Sumatriptan; Other: Placebo

INTERVENTIONS:
Drug: Sumatriptan — Single subcutaneous injection sumatriptan 6mg (in 0.5ml) in recovery
Other: Placebo — Single injection saline 0.5ml subcutaneously in recovery

SUMMARY:
Postoperative migrainous headache following craniotomy is distressing and may cause significant morbidity and often delay discharge from the hospital. The mechanism of this post craniotomy migraine is multifactorial. Possible causes include the intraoperative loss of cerebrospinal fluid leading to stretching of the dura, traction on intracranial vessels and meningeal irritation. There are two groups of patients who undergo elective minimally invasive craniotomies and yet have considerable postoperative migraine headache postoperatively. These are patients who have a craniotomy for clipping of an unruptured cerebral aneurysm and patients who require a microvascular decompressive craniotomy for cranial nerve pain such as trigeminal neuralgia. Their postoperative migrainous headache often impairs the quality of their recovery and may even delay discharge from hospital. Opioid analgesics are not always effective and may also worsen the postoperative nausea and vomiting and in turn postoperative quality of their recovery. Sumatriptan is a drug that has been used for decades for the treatment of migraine headaches. It acts on 5hydroxytryptophan receptors, which are located in the dura mater (lining of the brain) and are also located around the cranial trigeminal nerve ganglion. Thus sumatriptan may be an effective to improve postoperative migraine , nausea and vomiting and overall quality of recovery. We plan to do a randomized double blind placebo controlled trial on the effect of Sumatriptan for postoperative migraine on the postoperative quality of recovery after elective minimally invasive craniotomies. A total of 92 patients scheduled to undergo minimally invasive craniotomy for either clipping of an unruptured aneurysm or microvascular decompression for cranial nerve neuralgias will be included in this study. Patients within the 2 surgical groups with postoperative migraine will then be block randomized to receive either 6mg of sumatriptan subcutaneously or placebo following assessment in the post operative care unit (PACU). The primary outcome measure will be quality of recovery at 24 hours using Quality of recovery 40 Questionnaire (QoR-40). Our secondary outcome will be postoperative pain, analgesic consumption, side effects and hospital discharge times.

DETAILED DESCRIPTION:
Recently there have been changes in the surgical management of many patients who have an unruptured cerebral aneurysm and or cranial nerve neuralgia pain. The surgical technique now consists of a minimally invasive craniotomy that is less invasive with a smaller incision, shorter duration of procedure and in some patients the possibility of going home the same day, Postoperative surgical pain from the incision itself is usually minimal and they are usually managed very well with combination of both opioid and non-opioid analgesics such as fentanyl, morphine, hydromorphone, codeine, oxycocet, oxycontin and acetaminophen. In addition, up to 65% patients undergoing craniotomy may suffer from post craniotomy headache and the incidence may be higher after posterior fossa craniotomy. (1) Patients often complain of severe migraine headache associated with photophobia, nausea and vomiting and general feeling of unwell. These discomforts often delay discharge from the hospital and affect the quality of recovery. (2,3) Post craniotomy surgical pain usually decreases significantly after 24 hours whereas post craniotomy migraine headache, which may be a separate entity, continues for a longer period of time. (4) This migraine headache is in different location from the surgical incision and the conventional treatments of post surgical pain are ineffective against migraine headache.(5) Hence these patients usually suffer a lot after minimally invasive craniotomy. The mechanisms of postoperative migraine are also poorly understood and may be multifactorial including raised intracranial pressure, traction on intracranial blood vessels or meningeal irritation. (6) These factors activate the trigeminal afferent C fibres that reside on pial and dural blood vessels. This causes transmission of pain and release of neurogenic peptides activating an inflammatory cascade causing vasodilation and perivascular inflammation. The loss of cerebrospinal fluid is another factor.(7) With a minimally invasive craniotomy, loss of cerebrospinal fluid is unavoidable as it is needed for better surgical access. Serotonin (5-hydroxytryptophan) is a neurotransmitter that is thought to contribute to the feeling of wellbeing. There are receptors for 5hydroxytryptophan (5-HT) located in the central nervous system especially in the trigeminal nerve both near the dura as well as in brainstem (near the trigeminal nuclei) and also located on vascular endothelium and smooth muscle in meningeal blood vessels as well as in neuronal tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having elective craniotomy for clipping of unruptured intracranial aneurysm
2. Patients having craniotomy and microvascular decompression for cranial nerve neuralgia
3. Age 18-80
4. ASA I -III

Exclusion Criteria:

1. Patients with a known history of hypersensitivity to Sumatriptan or sulphonamides
2. Patients with a known history of Migraine
3. Patients who is on regular treatment with Sumatriptan
4. Patients with history of Ischemic heart disease - Angina, Myocardial infarction.
5. Patients who had rupture of their intracranial aneurysm.
6. Patients with history of severe liver disease.
7. Patients with history of stroke or uncontrolled hypertension
8. Inability to give informed consent
9. Pregnant patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2019-10-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery | 24 hours
  Using the validated Quality of Recovery 40 Questionnaire (QoR-40)

SECONDARY OUTCOMES:
Post operative pain scores | 24 hours
  Surgical site pain scores reported in the PACU. The numeric rating scale (NRS 0-10; 0, no pain; 10, worst pain imaginable) validated for measuring postoperative pain intensity. This scale is often used to divide patients into groups who are in need of pain treatment (moderate and severe pain) and those who are not (mild pain).
Post operative headache scores | 24 hours
  The Migraine-Specific Symptoms and Disability criteria and the Migraine Headache Index are used to characterize migraine symptoms in patient population before and after decompressive surgery.
Total analgesic consumption | 24 hours
  Postoperative analgesic consumption will be assessed in the two groups
Time to first opioid administration | less than 24 hours
  Monitoring the time of the first opioid dose in recovery room
Postoperative nausea and vomiting | less than 24 hours
  The incidence of PONV throughout the postoperative period
Hospital discharge time | less than one week
  Time to hospital discharge is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Lashmi Venkatraghavan, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Venkatraghavan L, Li L, Bailey T, Manninen PH, Tymianski M. Sumatriptan improves postoperative quality of recovery and reduces postcraniotomy headache after cranial nerve decompression. Br J Anaesth. 2016 Jul;117(1):73-9. doi: 10.1093/bja/aew152. PMID 27317706